CLINICAL TRIAL: NCT06507293
Title: Comparison of the Effects of Paravertebral Block and Erector Spinae Plane Block on Intraoperative Opioid Consumption Using NoL Index in Thoracotomy
Brief Title: Paravertebral Block and Erector Spinae Plane Block on Intraoperative Opioid Consumption Using NoL Index
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hadi Ufuk Yörükoğlu, Principal investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KAD-FR-01
Record Dates: First submitted 2024-07-01; First posted 2024-07-18 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain; Opioid Use
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP Group (Active Comparator): Patients who will receive erector spinae plane block
  Interventions: Procedure: Erector spiane plane block
- PVB Group (Active Comparator): Patients who will receive paravertebral block
  Interventions: Procedure: Paravertebral block

INTERVENTIONS:
Procedure: Paravertebral block — Before the general anesthesia induction, paravertebral block will be performed at T5 with 0.25% bupivacaine (20 mL) using ultrasound.
  Arms: PVB Group
Procedure: Erector spiane plane block — Before the general anesthesia induction, erector spinae plane block will be performed at T5 with 0.25% bupivacaine (20 mL) using ultrasound.
  Arms: ESP Group

SUMMARY:
Thoracotomy is among the most painful surgical procedures and can cause severe pain with a high incidence. Inadequate treatment of acute postoperative pain may lead to undesired complications. Paravertebral block (PVB) is an effective technique that provides adequate analgesia in thoracic surgeries. However, it is an advanced technique with potential complication risks. Erector spinae plane block (ESPB) is a relatively new and considered as a safer technique that provides comparable analgesia. However, the results are controversial and there are few studies that compares the effect of these blocks in thoracic surgeries. As well as the undesired effects of inadequate pain management, high doses of perioperative opioid usage may contribute to the development of dose-dependent long-term adverse events. Hemodynamic parameters are generally used to determine the intraoperative need for opioids in patients; however, hemodynamic parameters are not standardized and they do not provide a clear assessment. The Nociception Level (NoL) index is generated from five different parameters (heart rate, heart Rrate variability, photo-plethysmographic waveform amplitude, skin conductance level, number of skin conductance fluctuations, and their time derivatives) using a finger probe and is a promising monitoring technique. Selecting an effective analgesia method and determining the appropriate dose of opioids using NoL monitoring can reduce perioperative and postoperative complications and shorten hospital stays, allowing patients to return to daily life sooner. Additionally, preventing chronic pain syndromes that may develop in patients with inadequate analgesia, personalizing each patient's analgesia level, reducing healthcare costs, and improving quality of life can be achieved. The data from this study can demonstrate the analgesic efficacy of simpler regional anesthesia techniques, contributing to the widespread adoption of regional anesthesia applications, which is a crucial step in multimodal analgesia, thereby ensuring more effective pain management for surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergo elective thoracotomy surgery
* ASA physical status I-III

Exclusion Criteria:

* Spinal deformities
* BMI>35
* Patiens <50 kg
* Allergies to study medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Remifentanil consumption | Intraoperative
  Total amount of remifentanil used during the surgery (mg)
NRS Scores | Postoperative 1st, 6th, 12th and 24th hours
  Numeric Rating Scale scores, between 0-10 (0= no pain, 10=worst pain imaginable)
Morphine consumption | Postoperative 1st, 6th, 12th and 24th hours
  Amount of morphine in the postoperative period (mg)

SECONDARY OUTCOMES:
Rescue analgesic | Postoperative 1st, 6th, 12th and 24th hours
  The use of rescue analgesic
Nausea and vomiting | Postoperative 1st, 6th, 12th and 24th hours
  If the patient had nausea or vomiting, it will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hadi Ufuk Yörükoğlu, Principal Investigator — Kocaeli University, Department of Anesthesiology and Reanimation
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No